CLINICAL TRIAL: NCT00228072
Title: Suction-Curettage vs. Standard Excision in Axillary Hyperhidrosis
Brief Title: Liposuction as Treatment for Excessive Axillary Sweat
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VF20030189
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Hyperhidrosis
Keywords: Hyperhidrosis; Axillary; Excision; Suction-curettage; Outcome
MeSH Terms: conditions — Hyperhidrosis | interventions — Vacuum Curettage

INTERVENTIONS:
Procedure: Suction-curettage

SUMMARY:
The purpose of this study is to determine if suction-curettage of the axilla is favorable in regard to effect, recovery and cosmetic appearance compared to standard surgical excision of the skin of the axilla in case of excessive sweating.

DETAILED DESCRIPTION:
The surgical standard treatment for isolated excessive axillary sweating is excision of the hair-bearing area of the axilla. This technique is associated with a risk of impaired wound healing, infections, wide scars and a risk of impairment in the movement of the arm (seldom).

A new technique suction-curettage, much alike the liposuction technique, in which the dermis is curettage from a sub-dermal approach with a cutting and sucking devise, may be promising in regard to recovery and cosmetic appearance postoperatively, but the effect of the sweat production is not well known. This study compares liposuction vs. standard excision in individuals with isolated excessive isolated axillary sweating randomized to treatment with one of each technique in both axillas.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals with primary axillary hyperhidrosis

Exclusion Criteria:

* Secondary axillary hyperhidrosis
* Hidrosadenitis axillaris/inguinalis
* Prior surgery
* Iontophoresis or botox treatment 12 months prior
* Known hypersensitivity to local analgetics (lidocaine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Primary Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Finn Gottrup, DMsci, Study Chair — University Center of Wound Healing, Dept. of Plastic Surgery, Odense University Hospital, Sdr. Boulevard 29, DK-5000 Odense C, Denmark; Torben Moeller-Christensen, MD, Study Director — Department of Plastic Surgery, Odense University Hospital, Sdr. Boulevard 29, DK-5000 Odense C, Denmark
Locations (1):
- Department of Plastic Surgery, Odense University Hospital, Odense, Fyn, Denmark